CLINICAL TRIAL: NCT03316248
Title: Investigation of the Effect of Visual Feedback on Function, Stability and Quality of Life in Individuals With Transtibial Amputation
Brief Title: The Effect of Visual Feedback on Function, Stability and Quality of Life in Transtibial Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Kırdı, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO 17 / 115
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Amputation; Traumatic Amputation
Keywords: Transtibial amputation; visual feedback; rehabilitation
MeSH Terms: conditions — Amputation, Traumatic | interventions — Feedback, Sensory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual feedback (Experimental): participants in the experimental group were applied usual prosthetic rehabilitation with visual feedback methods. 9 sessions for three days were applied.
  Interventions: Other: visual feedback
- Usual prosthetic rehabilitation (Active Comparator): participants in the control group were applied usual prosthetic rehabilitation. 9 sessions for three days were applied.
  Interventions: Other: usual prosthetic rehabilitation

INTERVENTIONS:
Other: visual feedback — in the study group, subjects were applied for example prosthetic weight bearing exercises in front of the mirror. They watched their reflected image while doing exercises.
  Arms: visual feedback
Other: usual prosthetic rehabilitation — prosthetic weight bearing and balance exercises were applied to the control group for 9 sessions.
  Arms: Usual prosthetic rehabilitation

SUMMARY:
This study was conducted to examine the effect of visual feedback on function, stability and quality of life in transtibial amputees. A total of 24 subjects who had unilateral transtibial amputations, used prosthesis with total surface bearing socket (TSB) for at least 1 year and volunteered to participate in the study were included. Before and after Treatment subjects were evaluated with "LASAR Posture" for prosthetic weight bearing (PWB), "Berg Balance Scale (BBS)" and "Timed Up& Go Test (TUG)" for balance and functional mobility, "2-Minute-Walk-Test (2MWT)" for physical performance, "Satisfaction with the Prosthesis Questionnaire (SATPRO)" for prosthetic pleasure and "Nottingham Health Profile (NHP)" for health- related quality of life. Participants were randomly divided into two equal groups as study and control groups. After the evaluations the same exercises; PWB exercises, balance exercises, anteroposterior and lateral weight shifting, obstacle course, walking on different grounds were applied to the the study group with visual feedback methods and control group.

DETAILED DESCRIPTION:
Inclusion criteria:

1. had transtibial amputation
2. >18 years old
3. had total surface bearing socket at least one year

Outcome measures:

* Prosthetic weight bearing
* Berg Balance Scale
* Timed up &go Test
* 2 Minute Walk Test
* Satisfaction of prosthesis questionnare
* Nottingham health profile

ELIGIBILITY:
Inclusion Criteria:

* had unilateral transtibial amputations,
* used prosthesis with total surface bearing socket (TSB) for at least 1 year
* volunteered to participate in the study

Exclusion Criteria:

* had any neurological disorders
* had any cognitive problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-06-18 (Actual)

PRIMARY OUTCOMES:
Prosthetic Weight bearing | 3 minutes
  minimal (Min WB) and maximal (Max WB) values were visually recorded on the amputated side for three consecutive minutes.
  The average weight bearing on the amputated side (Ml) was calculated by dividing the sum of maximal and minimal weight bearing values by two.
  The percentage of total body weight (TBW) borne through the amputated limb was then determined using the formula:
  (Ml/TBW) x 100

CONTACTS AND LOCATIONS:
Overall Officials: Elif Kırdı, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No